CLINICAL TRIAL: NCT02243176
Title: SMART Study - A 24-Week, Multicenter, Randomized, Parallel-group, Open-label, Active Controlled Phase IV Study to Assess the Efficacy, Safety and Tolerability of Saxagliptin Compared With Acarbose When in Combination With Metformin in Patients With Type 2 Diabetes Mellitus (T2D) Inadequately Controlled With Metformin Monotherapy
Brief Title: 24-Week, Multicenter, Randomized, Parallel-group, Open-label, Active Controlled Phase IV Study to Assess the Efficacy, Safety and Tolerability of Saxagliptin Compared With Acarbose When in Combination With Metformin in Patients With T2D Inadequately Controlled With Metformin Monotherapy
Acronym: SMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1680L00018
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Saxagliptin; Acarbose; Type 2 Diabetes; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin (Experimental): The dose of saxaglitpin will be 5mg oral qd. An estimated total of 480 patients (240 per treatment arm) will be randomized in a 1:1 ratio to the active treatment arm and the active comparator arm. So estimated 240 patients will be allocated to this arm.
  Interventions: Drug: Saxagliptin
- Acarbose (Active Comparator): Patients who take acarbose will begin with 50mg tid for 7 days then be titrated to 100mg tid till the end of the study. A call visit (V5) will be performed at Week 1 for adverse event and reminding patients the dose titration of acrabose. An estimated total of 480 patients (240 per treatment arm) will be randomized in a 1:1 ratio to the active treatment arm and the active comparator arm. So estimated 240 patients will be allocalted to this arm.
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Saxagliptin — The dose of saxaglitpin will be 5mg oral qd.
  Other Names: Onglyza
  Arms: Saxagliptin
Drug: Acarbose — Patients who take acarbose will begin with 50mg tid for 7 days then be titrated to 100mg tid till the end of the study. A call visit (V5) will be performed at Week 1 for adverse event and reminding patients the dose titration of acrabose.
  Other Names: Glucobay
  Arms: Acarbose

SUMMARY:
SMART Study - A 24-Week, Multicenter, Randomized, Parallel-group, Open-label, Active Controlled Phase IV Study to Assess the Efficacy, Safety and Tolerability of Saxagliptin Compared with Acarbose when in Combination with Metformin in Patients with Type 2 Diabetes Mellitus (T2D) Inadequately Controlled with Metformin Monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes mellitus
2. Men and women (non-pregnant and using a medically approved birth-control method) aged at least 18 years at screening.
3. T2D patients treated with stable metformin monotherapy for at least 8 weeks prior to screening. Metformin dose should be ≥ 1500 mg/day (or individual maximally tolerated dose), but not more than the maximum dose specified in the label
4. HbA1c ≥ 7.5% and ≤ 11.0% at screening or within 4 weeks prior to screening (by local laboratory) and HbA1c ≥ 7.0% and ≤ 11.0% at pre-randomization visit (by central laboratory)
5. FPG ≤ 13.3 mmol/L (≤ 240 mg/dL) at pre-randomization visit (by central laboratory)
6. Able and willing to provide written informed consent and to comply with the study protocol

Exclusion Criteria:

1. Women who are pregnant, intending to become pregnant during the study period, lactating females, or women of child-bearing potential not using highly effective, medically approved birth control methods.
2. Diagnosis or history of:

   1. Type 1 diabetes mellitus, diabetes resulting from pancreatic injury or secondary forms of diabetes, eg, acromegaly or Cushing's syndrome.
   2. Acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma within the past 6 months.
3. Previous treatment with any dipeptidyl peptidase-4 (DPP4) inhibitor or GLP-1 receptor agonists within the past one year.
4. History of hypersensitivity reaction (e.g., anaphylaxis, angioedema, exfoliative skin conditions) to dipeptidyl peptidase-4 inhibitor (DPP4) or Acarbose.
5. Treatment with any anti-diabetic medication for more than 7 consecutive days other than metformin in the last 8 weeks prior to screening

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Shanghai, China

REFERENCES:
- [Derived] Du J, Liang L, Fang H, Xu F, Li W, Shen L, Wang X, Xu C, Bian F, Mu Y. Efficacy and safety of saxagliptin compared with acarbose in Chinese patients with type 2 diabetes mellitus uncontrolled on metformin monotherapy: Results of a Phase IV open-label randomized controlled study (the SMART study). Diabetes Obes Metab. 2017 Nov;19(11):1513-1520. doi: 10.1111/dom.12942. Epub 2017 Jul 6. PMID 28296055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 689 patients were enrolled into this study from 35 sites in China. The enrolled patient number ranged from 10 to 58 among 24 centers, and 2 to 9 patients from eight centers, none was enrolled in 3 centers. The enrolment period was from 24 Sep 2014 to 29 Sep 2015.
Pre-assignment Details: A total of 201 patients were enrolled but not randomized: 171 patients did not meet eligibility criteria, and 24 patients were voluntary discontinuations, two patients developed study-specific withdrawal criteria, one patient lost follow-up, and three patient failed due to other reasons
Period: Overall Study
Arm/Group | Saxagliptin | Acarbose
Started | 244 (3 of the randomized subjects withdrew before taking any medication) | 244
Completed | 230 | 229
Not Completed | 14 | 15
Not completed — Other reason | 1 | 2
Not completed — protocol specified withdrawal critera | 1 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Full analysis set included all randomized subjects who took at least 1 randomized IP dose, and had at least 1 non-missing baseline and 1 post-baseline efficacy data assessments
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin | Acarbose | Total
Number analyzed (Participants) | 238 | 243 | 481
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (10.51) | 56.5 (10.81) | 55.6 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 105 | 196
  Male | 147 | 138 | 285
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (China Mainland) | 238 | 243 | 481
Height [Mean (Standard Deviation); unit: cm] | 166.3 (8) | 165.9 (7.75) | 166.1 (7.87)
Weight [Mean (Standard Deviation); unit: kg] | 73.3 (12.61) | 72.6 (12.27) | 72.9 (12.43)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 26.4 (3.47) | 26.3 (3.49) | 26.3 (3.48)
Duration of diabetes mellitus (years) [Mean (Standard Deviation); unit: Years] | 5.1 (4.4) | 5.3 (4.76) | 5.2 (4.58)
Type of diabetes mellitus [Number; unit: Participants]
  Type 2 | 238 | 243 | 481
  Other | 0 | 0 | 0
Currently taking antidiabetic medication [Number; unit: Participants] | 238 | 243 | 481
Any diabetes mellitus complications [Number; unit: Participants]
  No | 214 | 221 | 435
  Yes | 24 | 22 | 46
Any relevant medical conditions [Number; unit: Participants]
  Yes | 119 | 125 | 244
  No | 65 | 64 | 129
  Missing | 54 | 54 | 108
Any current medication，excluding antidiabetic drugs [Number; unit: Participants]
  Yes | 59 | 73 | 132
  No | 179 | 170 | 349
HbA1c (%) [Mean (Standard Deviation); unit: %] — Haemoglobin A1c
  % | 8.23 (0.85) | 8.16 (0.81) | 8.20 (0.83)
FPG [Mean (Standard Deviation); unit: mmol/l] — Fasting Plasma Glucose
  mmol/l | 9.01 (2.14) | 8.81 (1.95) | 8.90 (2.04)
2hPPG [Mean (Standard Deviation); unit: mmol/l] — 2h Postprandial Plasma Glucose
  mmol/l | 11.17 (2.82) | 10.25 (2.89) | 10.7 (2.89)
Triglycerides [Mean (Standard Deviation); unit: mmol/l] | 1.99 (1.12) | 1.96 (1.38) | 1.97 (1.26)
TC [Mean (Standard Deviation); unit: mmol/l] — Total Cholesterol
  mmol/l | 4.78 (1.07) | 4.82 (0.94) | 4.80 (1.01)
LDL [Mean (Standard Deviation); unit: mmol/l] — Low Density Lipoprotein-Cholesterol
  mmol/l | 2.73 (0.89) | 2.77 (0.79) | 2.75 (0.84)
HDL [Mean (Standard Deviation); unit: mmol/l] — High Density Lipoprotein-Cholesterol
  mmol/l | 1.16 (0.29) | 1.2 (0.3) | 1.18 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in HbA1c at Week 24 (DAO)
Description: Primary Objective: Efficacy of saxagliptin plus metformin on glycemic control compared with acarbose plus metformin in patients with T2D inadequately controlled with metformin. By Measure absolute change from baseline in HbA1c at Week 24
Time Frame: From baseline to 24 week
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: % (HbA1c)
Arm/Group | Saxagliptin | Acarbose
Number analyzed (Participants) | 238 | 243
% (HbA1c) | -0.82 (0.06) | -0.78 (0.06)
Statistical Analysis 1: Comparison: Saxagliptin vs Acarbose; H01: μS-μA≥ 0.4% vs Ha1: μS-μA< 0.4%. Null hypothesis will be rejected if the upper limit of 2-sided 95% CI is below 0.4%.If the null hypothesis above (H01) is rejected, the following hypothesis will be tested to further establish superiority: H02: μS-μA≥ 0 vs Ha2: μS-μA< 0. This null hypothesis (H02) will be rejected if the upper limit of 2-sided 95% CI is below 0; Test type: Non-Inferiority or Equivalence — With a total sample size of 480 patients randomized and an expected drop-out rate of 20%, the trial will be powered at 90% to establish non-inferiority for the primary endpoint, at a one-sided alpha level of 0.025, with the non-inferiority margin of 0.4%, assuming the true effects are the same between treatments. The calculation is also based on the assumption that the standard deviation for the change in HbA1c is 1.2%; p = 0.6236, Mixed Model Repeated Measures — This p value is for the hypothesis of superiority; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.22 to 0.13], Standard Error of Mean 0.09 — Mean difference=Saxagliptin - Acarbose

2. Primary Outcome: Absolute Change From Baseline in HbA1c at Week 24 (DAO)
Description: The primary endpoint was analyzed based on Per protocol analysis set as the supportive analysis.
Time Frame: From baseline to 24 week
Population: The Per Protocol analysis set was a subset of the Full analysis set that included subjects who did not have significant protocol deviations that affect the study outcome. The exclusions from the PP analysis set was determined prior to database lock.
Measure: Least Squares Mean (Standard Error); unit: % (HbA1c)
Arm/Group | Saxagliptin | Acarbose
Number analyzed (Participants) | 219 | 204
% (HbA1c) | -0.83 (0.06) | -0.80 (0.07)
Statistical Analysis 1: Comparison: Saxagliptin vs Acarbose; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7809, Mixed Model Repeated Measures — This p value is for the hypothesis of superiority; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.21 to 0.15], Standard Error of Mean 0.09 — Mean difference=Saxagliptin - Acarbose

3. Secondary Outcome: Proportion (%) of Patients With Any GI Adverse Events
Description: Secondary Objective: Assessment of any gastrointestinal adverse events of saxagliptin versus acarbose. by measure proportion (%) of patients with any gastrointestinal adverse events.
Time Frame: 24 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Saxagliptin | Acarbose
Number analyzed (Participants) | 238 | 243
percentage of participants
  NO | 94.5 | 75.3
  YES | 5.5 | 24.7
Statistical Analysis 1: Comparison: Saxagliptin vs Acarbose; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratefied by the baseline disease severity (HbA1c < 8.0% and ≥ 8.0%); Risk Ratio (RR) = 0.22, 95% CI 2-sided [0.12 to 0.39] — RR = Saxagliptin/Acarbose

4. Secondary Outcome: Proportion (%) of Patients Achieving a Therapeutic Glycemic Response Defined as HbA1c<7.0%
Description: Secondary Objective: Effects of saxagliptin versus acarbose on the additional parameters, by measure proportion (%) of patients achieving a therapeutic glycemic response defined as HbA1c<7.0%
Time Frame: 24 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Saxagliptin | Acarbose
Number analyzed (Participants) | 230 | 229
percentage of participants | 38.3 | 41.5
Statistical Analysis 1: Comparison: Saxagliptin vs Acarbose; Test type: Superiority or Other; p = 0.5044, Cochran-Mantel-Haenszel; stratefied by baseline disease severity (HbA1c<8%, >=8%); Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.74 to 1.15]

5. Secondary Outcome: Proportion (%) of Patients Achieving HbA1c<7.0% Without GI Adverse Events
Description: Secondary Objective: Assessment of any gastrointestinal adverse events of saxagliptin versus acarbose. by measure proportion (%) of patients achieving HbA1c<7.0% without GI adverse events.
Time Frame: Whole study duration
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Saxagliptin | Acarbose
Number analyzed (Participants) | 230 | 229
percentage of participants | 37.0 | 28.8
Statistical Analysis 1: Comparison: Saxagliptin vs Acarbose; Test type: Superiority or Other; p = 0.0518, Cochran-Mantel-Haenszel; Stratefied by the baseline disease severity (HbA1c < 8.0% and ≥ 8.0%); Risk Ratio (RR) = 1.28, 95% CI 2-sided [0.98 to 1.67] — RR = Saxagliptin/Acarbose

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Secondary objective: Effects of saxagliptin versus acarbose on the additional parameters, by measure change from baseline in fasting plasma glucose, 2h postprandial glucose, β-cell function, body weight at week 24
Time Frame: From baseline to 24 week
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mmol/l
Arm/Group | Saxagliptin | Acarbose
Number analyzed (Participants) | 238 | 243
mmol/l | -0.99 (0.13) | -1.01 (0.13)
Statistical Analysis 1: Comparison: Saxagliptin vs Acarbose; Test type: Superiority or Other; p = 0.8915, Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.33 to 0.38], Standard Error of Mean 0.18 — Mean difference=Saxagliptin - Acarbose

7. Secondary Outcome: Change From Baseline in 2H Postprandial Glucose (2HPPG)
Description: as for outcome 6
Time Frame: From baseline to 24 week
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mmol/l
Arm/Group | Saxagliptin | Acarbose
Number analyzed (Participants) | 227 | 232
mmol/l | -0.77 (0.176) | -1.07 (0.174)
Statistical Analysis 1: Comparison: Saxagliptin vs Acarbose; Test type: Superiority or Other; p = 0.2248, ANCOVA; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.186 to 0.791], Standard Error of Mean 0.249 — Mean difference=Saxagliptin - Acarbose

8. Secondary Outcome: Change From Baseline in HOMA-β
Description: Secondary objective: Effects of saxagliptin versus acarbose on the additional parameters, by measure change from baseline in fasting plasma glucose, 2h postprandial glucose, β-cell function was estimated by the Homeostasis model assessment-β (HOMA-β), which was defined as fasting insulin (mU/mL) x 20 / (fasting glucose (mmol/mL) - 3.5, body weight at week 24
Time Frame: From baseline to 24 week
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: mU/mmol
Arm/Group | Saxagliptin | Acarbose
Number analyzed (Participants) | 227 | 225
mU/mmol | 20.56 (5.932) | 13.08 (5.958)
Statistical Analysis 1: Comparison: Saxagliptin vs Acarbose; Test type: Superiority or Other; p = 0.3739, ANCOVA; Mean Difference (Final Values) = 7.48, 95% CI 2-sided [-9.039 to 24.005], Standard Error of Mean 8.407 — Mean difference=Saxagliptin - Acarbose

9. Secondary Outcome: Change From Baseline in Body Weight
Description: as for outcome 6
Time Frame: From baseline to 24 week
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Saxagliptin | Acarbose
Number analyzed (Participants) | 238 | 243
kg | -1.36 (0.18) | -2.05 (0.18)
Statistical Analysis 1: Comparison: Saxagliptin vs Acarbose; Test type: Superiority or Other; p = 0.0078, Mixed Model Repeated Measures; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [0.18 to 1.19], Standard Error of Mean 0.26 — Mean difference=Saxagliptin - Acarbose

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from time of signature of informed consent, throughout the treatment period. That was about 28 weeks for every subject.
Description: Unresolved AEs unresolved at the subject's last visit were followed up by the Investigator for as long as medically indicated, but without furtherrecording in the CRF. Below reported AEs were Treatment Emergent Adverse Events which were AEs from the first dose of investigational product to the end of follow-up.
Arm/Group | Saxagliptin | Acarbose
Serious Adverse Events (participants affected / at risk) | 5/241 | 2/244
Other Adverse Events (participants affected / at risk) | 27/241 | 74/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saxagliptin (N=241) | Acarbose (N=244)
herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) — The SOC term was reported as "General disorders and administration site conditions" in study results.
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saxagliptin (N=241) | Acarbose (N=244)
Hyperlipidaemia (Metabolism and nutrition disorders) | 15 (15) | 14 (14)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (9) | 17 (17)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 25 (25)
Flatulence (Gastrointestinal disorders) | 0 (0) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days